CLINICAL TRIAL: NCT04348136
Title: An Extension Study of JR-141 in Patients With Mucopolysaccharidosis Type II
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-141-302
Record Dates: First submitted 2019-12-18; First posted 2020-04-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JR-141 (Experimental)
  Interventions: Drug: JR-141

INTERVENTIONS:
Drug: JR-141 — IV infusion, 2.0 mg/kg/week

SUMMARY:
Multicenter, open-label, single-group, designed to evaluate the long term efficacy and safety of study drug for the treatment of the MPS II.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who participated in the preceding Study JR-141-301 and completed the Week 52 visit, and has no safety concerns to enter this study in the opinion of the investigator or subinvestigator.
2. A patient capable of providing written informed consent in person (However, this is not required for patients aged younger than 20 years at the time of consent or patients with intellectual disability associated with MPS II whose willingness cannot be verified.)
3. For patients aged younger than 20 years at the time of consent or patients with intellectual disability associated with MPS II whose willingness cannot be verified, written consent must be obtained from the legally acceptable representative. (Wherever possible, written consent of the patient should be obtained.)
4. Male patient whose partner is of child-bearing potential and agrees to use a medically accepted, highly effective method of contraception.

Exclusion Criteria:

1. A patient who used any concomitant medication or therapy that could affect study assessments in the opinion of the investigator or subinvestigator.
2. A patient with a history of serious drug allergy or hypersensitivity that precludes participation in this study in the opinion of the investigator or subinvestigator.
3. A patient judged to be ineligible by the investigator or subinvestigator for other reasons.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | From the start of study (Week 52 of preceding study) up to the end of study, up to approximately 10.6 years
Occurrence of adverse reactions | From the start of study (Week 52 of preceding study) up to the end of study, up to approximately 10.6 years
Incidence of abnormal vital signs | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
  Laboratory tests (hematology)
Incidence of abnormal vital signs | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
  Laboratory tests (biochemistry)
Incidence of abnormal vital signs | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
  Laboratory tests (iron-related tests)
Laboratory tests (urinalysis) | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Vital signs (pulse rate) | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Vital signs (body temperature) | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Vital signs (blood pressure) | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
12-lead electrocardiogram | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
  The presence or absence of abnormal findings (if present, specific findings and whether or not they are reported as adverse events)
Antibody tests (anti-JR-141 antibodies) | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
IAR | From the start of study (Week 52 of preceding study) up to the end of study, up to approximately 10.6 years
Time course of developmental assessment data (Kyoto Scale of Psychological Development 2001) from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of developmental assessment data (Vineland-II) from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of developmental assessment data (Bayley-III or KABC-II) from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of CSF substrate (HS and DS) concentrations from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of serum HS and DS concentrations from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of urinary HS concentration from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of urinary DS concentration from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of uronic acid concentration from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of liver volume (assessed by CT or MRI) from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of spleen volume (assessed by CT or MRI) from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of cardiac function (assessed by echocardiography) from initial dosing in the preceding study | Week 78, 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of 6-minute walk test distance from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years
Time course of joint range of motion from initial dosing in the preceding study | Week 104, an average of 52 weeks after Week 104, up to approximately 10.6 years

CONTACTS AND LOCATIONS:
Locations (20):
- Japan (20):
  - Fukui Clinical site, Fukui
  - Fukuoka Clinical site 2, Fukuoka
  - Fukuoka Clinical site, Fukuoka
  - Gifu Clinical site, Gifu
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hokkaido Clinical site, Hokkaido
  - Kananagawa Ckinical site, Kanagawa
  - Kumamoto Clinical site, Kumamoto
  - Okayama Clinical site, Okayama
  - Okayama Clinical site 2, Okayama
  - Okinawa Clinical site, Okinawa
  - Osaka Clinical site 3, Osaka
  - Osaka Clinical site 2, Osaka
  - Osaka Clinical site, Osaka
  - Saitama Clinical site, Saitama
  - Shizuoka Clinical site, Shizuoka
  - Shizuoka Clinical site 2, Shizuoka
  - Tochigi Clinical site, Tochigi
  - Tokyo Clinical site, Tokyo
  - Tottori Clinical site, Tottori